CLINICAL TRIAL: NCT06397976
Title: The Heidelberg Engineering ANTERION Software Comparison Precision and Agreement Study
Status: Terminated | Type: Observational
Why Stopped: newer version of the devices available for testing
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B-2023-2
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-11

CONDITIONS: Eyes With Normal Anterior Segment; Eyes With Abnormal Anterior Segment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Eyes with normal anterior segment
  Interventions: Device: ANTERION investigational
- Eyes with abnormal anterior segment
  Interventions: Device: ANTERION investigational

INTERVENTIONS:
Device: ANTERION investigational — Measurements from the investigational device ANTERION with software version 1.5 are to be compared against measurements from the ANTERION with software version 1.2.4 (cleared version)

SUMMARY:
This study is conducted to compare the the investigational device ANTERION with software version 1.5 against the ANTERION with software version 1.2.4 (cleared version)

ELIGIBILITY:
Inclusion Criteria Normal Anterior Segment

1. Age 22 years or older
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions
3. Able to fixate
4. Eye(s) with normal anterior segment

Exclusion Criteria Normal Anterior Segment

1. Active infection or inflammation in the study eye
2. Insufficient tear film or corneal reflex
3. Physical inability to be properly positioned at the study devices or eye exam equipment
4. Rigid contact lens wear 2 weeks prior to imaging
5. Soft lenses worn within one hour prior to imaging
6. Cataract grade ≥1.5

Inclusion Criteria Abnormal Anterior Segment

1. Age 22 years or older
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions
3. Able to fixate
4. Eye(s) with abnormal anterior segment (including cataract grade ≥ 1.5)

Exclusion Criteria Abnormal Anterior Segment

1. Active infection or inflammation in the study eye
2. Insufficient tear film or corneal reflex
3. Physical inability to be properly positioned at the study devices or eye exam equipment
4. Rigid contact lens wear 2 weeks prior to imaging
5. Soft lenses worn within one hour prior to imaging

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eyes with normal and eyes with abnormal anterior segment population
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Central Cornea Thickness | Through study completion, an average of 1 day
  Reproducibility and repeatability of Central Cornea Thickness of ANTERION and the reference device
Thinnest Point Thickness | Through study completion, an average of 1 day
  Reproducibility and repeatability of Thinnest Point Thickness of ANTERION and the reference device
Lens Thickness | Through study completion, an average of 1 day
  Reproducibility and repeatability of Lens Thickness of ANTERION and the reference device
Anterior Chamber Depth | Through study completion, an average of 1 day
  Reproducibility and repeatability of Anterior Chamber Depth of ANTERION and the reference device
Axial Length | Through study completion, an average of 1 day
  Reproducibility and repeatability of Axial Length of ANTERION and the reference device

SECONDARY OUTCOMES:
Adverse Events Rate | Through study completion, an average of 1 day
  Adverse events found during the clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fischer, MD, Principal Investigator — Fischer Laser Eye Center
Locations (1):
- Fischer Eye Laser Center, Willmar, Minnesota, United States